CLINICAL TRIAL: NCT03344705
Title: Safety and Efficacy Evaluation of IM19 Chimeric Antigen Receptor-modified T Cells (IM19CAR-T) In CD19+ B Cell Malignancies
Brief Title: Safety and Efficacy Evaluation of IM19 Cells
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YMCART201701
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IM19 CART (Experimental): All patients will be treated with fludarabine and cyclophosphamide for 3 days,then,CAR-T cells expressing CD19 CAR will be infused 24-96 hours later.
  Interventions: Biological: IM19 CAR-T; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: IM19 CAR-T — All patients will be treated with fludarabine and cyclophosphamide for 3 days. Two days later, Cells Expressing an Anti-CD19 Chimeric Antigen Receptor will be infused.
  Other Names: IM19
Drug: Fludarabine — Two days before cell infusion,all patients will be treated with fludarabine for 3 days
  Other Names: F
Drug: Cyclophosphamide — Two days before cell infusion,all patients will be treated with cyclophosphamide for 3 days
  Other Names: C

SUMMARY:
Assessment of the Safety and Feasibility of Administering T cells Expressing an Anti-CD19 Chimeric Antigen Receptor to Patients With CD19+ B-cell Hematological Malignancies.

DETAILED DESCRIPTION:
Assessment of the Safety and Feasibility of Administering T cells Expressing an Anti-CD19 Chimeric Antigen Receptor to Patients With CD19+ B-cell Hematological Malignancies(including B-cell Acute lymphoblastic Leukemia、B-cell Chronic Lymphocytic Leukemia、Non-Hodgkin's lymphoma) and Determine the Best Dosage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CD19 positive relapsed or refractory B-cell malignancies, including B-cell Acute Lymphocytic Leukemia(ALL)、B-cell Chronic Lymphocytic Leukemia(CLL)、Non-Hodgkin's lymphoma(NHL).

1)Patients with ALL:

* Previously treated with at least two courses of chemotherapy Ⅱ The interval of the last chemotherapy and disease progression is less than one year.

  Ⅲ Not suitable for allogeneic stem cell transplantation. 2)Patients with CLL:
* Previously treated with at least two courses of chemotherapy

  Ⅱ The interval of the last chemotherapy and disease progression is less than two years.

  Ⅲ Not suitable for allogeneic stem cell transplantation conditions or due to conditions to abandon allogeneic stem cell transplantation.

  3) Patients with DLBCL or FL、PMBCL:
* Patients who relapsed or were refractory after at least two previous treatments.

  Ⅱ Patients who relapsed after transplantation. 4)Patients who have relapsed or have refractory mantle cell lymphoma after at least one treatment.

  2.Measurable disease,including minimal residual disease. 3.Gender is not limited, to be aged 4 to 75 years 4.Expected survival >3 months. 5.Eastern Cooperative Oncology Group(ECOG) score 0-2. 6.Women of childbearing potential must have a blood pregnancy test taken and proven negative prior to the treatment. All patients agree to use reliable methods of contraception during the trial period and until follow-up for the last time.

  7.Absence of symptoms of central nervous system(CNS) leukemia.

Exclusion Criteria:

1. Patients who have been treated with chemotherapy or radiotherapy within 2 weeks before blood collection.
2. Patients have GVHD, which needs treatment with immunosuppressive agents,or patients with autoimmune diseases.
3. Patient who have been treated with systemic steroid medication within two weeks of blood collection（Except for the recent or current use of inhaled steroids）.
4. Patient who have been treated with stimulation of bone marrow hematopoietic cells generated drugs(Such as Recombinant Human Granulocyte Colony-stimulating Factor Injection) within 2 weeks before the blood collection period to use .
5. The number of T cells in peripheral blood is lower than 2×10^8/L.
6. Previously treatment with any gene therapy products.
7. History of epilepsy or other CNS disease.
8. New York Heart Association(NYHA) grade≥Ⅲ.
9. Creatinine> 1.5×normal value，Alanine transaminase(ALT) /Aspartate aminotransferase(AST)>3×normal value，Bilirubin >2×normal value.
10. Degree of myeloproliferation： Ⅳ-V
11. Active hepatitis B , hepatitis C or HIV infection and cytomegalovirus infection ,Epstein-Barr virus infection or any other uncontrolled active infection.
12. Pregnancy or breast-feeding women.
13. Any uncontrolled medical disorders that the researchers considered are not suitable to participate the clinical trial.
14. Any situation that would increase dangerousness of subjects or disturb the outcome of the clinical study according to the researcher's evaluation.

Ages: 4 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-08-21 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events | 2 years
  defined as >= Grade 3 signs/symptoms,laboratory toxicities,and clinical events that are possibly,likely,or definitely related to study treatment Adverse events assessed according to NCI-CTCAE v4.0 criteria 2.

SECONDARY OUTCOMES:
Overall response rate | 2 years
  2. Overall response rate An objective response is defined as: (1) a morphologic complete response (CR) or (2) a complete response with incomplete recovery of counts (CRi) (based on NCCN guidelines (National Comprehensive Cancer Network (NCCN), 2014) or (3) a negative minimal residual disease assessed by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Hongmei Jing, MD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Bao F, Wan W, He T, Qi F, Liu G, Hu K, Lu XA, Yang P, Dong F, Wang J, Jing H. Autologous CD19-directed chimeric antigen receptor-T cell is an effective and safe treatment to refractory or relapsed diffuse large B-cell lymphoma. Cancer Gene Ther. 2019 Jul;26(7-8):248-255. doi: 10.1038/s41417-018-0073-7. Epub 2019 Jan 9. PMID 30622321